CLINICAL TRIAL: NCT05109949
Title: Acute Effect of Empagliflozin vs Dapagliflozin vs Placebo Administration Over Pulse Wave Velocity in Patients With Type Two Diabetes
Brief Title: Acute Effect of Empagliflozin vs Dapagliflozin Over Pulse Wave Velocity in Type Two Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Principal Investigator, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CUCS-INTEC-XOLOTL
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus Type 2 Without Complication
MeSH Terms: interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapagliflozin 10 mg (Experimental): Dapagliflozin is an oral medication used to treat Type 2 diabetes. It belongs to a sodium-glucose cotransporter 2 (SGLT2) inhibitors.
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Empagliflozin 25 mg (Experimental): Empagliflozin is an oral medication used to treat Type 2 diabetes. It belongs to sodium-glucose cotransporter 2 (SGLT2) inhibitors.
  Interventions: Drug: Empagliflozin 25 MG
- Placebo (Placebo Comparator): Calcinated magnesium is a white powdery compound, MgO, used in pharmaceuticals as binder.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Daily morning dose per oral of Dapagliflozin 10 mg for 7 days
  Other Names: Farxiga, Forxiga
  Arms: Dapagliflozin 10 mg
Drug: Empagliflozin 25 MG — Daily morning dose per oral of Empagliflozine 25 mg for 7 days
  Other Names: Jardiance
  Arms: Empagliflozin 25 mg
Other: Placebo — Daily morning dose per oral of Calcined magnesite 500 mg for 7 days
  Arms: Placebo

SUMMARY:
To date one of the main independent biomarkers of cardiovascular disease is the arterial stiffness parameters measured by carotid-femoral pulse wave velocity. It is known that SGLT2 inhibitors develop cardiac protection over long term administration, but there's not enough studies about acute effects in early administration.

DETAILED DESCRIPTION:
Measure basal carotid-femoral Pulse Wave Velocity through a Pulse Pen tonometer by DiaTecne among basic physical examination, blood test, anthropometric and hemodynamic measurements; then administrate randomly dapagliflozin 10 mg, empagliflozin 25 mg or placebo for 7 days and then perform all of the measurements and blood test again.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM
* HbA1c > 7 y < 10
* BMI 25 - 34.9 kg/m2
* Signature of consent under information

Exclusion Criteria:

* Hypertension
* Treated with insulin and / or loop diuretics and thiazides
* T1DM
* Hypotension
* Any autoimmune disease
* Liver disease
* Women whitout birth control method
* Women taking oral birth control or under hormone replacement therapy
* Woman pregnant or breastfeeding
* Untreated thyroid disease
* Patients with a cardiovascular disease that contraindicates the use of this pharmacological class
* Glomerular filtration rate <60ml/min (Cockcroft-Gault)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | 7 days
  Change from baseline carotid-femoral pulse wave velocity at 7 days. Using a PulsePen tonometer by DiaTechne.

SECONDARY OUTCOMES:
Fasting plasma glucose | 7 days
  Change from baseline, using the BioSystems® Glucose Oxidase / Peroxidase kit; in an automated clinical chemistry analysis equipment brand XL-100Erba
Total cholesterol | 7 days
  Change from baseline, using the BioSystems® Glucose Oxidase / Peroxidase kit.
Triglycerides | 7 days
  Change from baseline, using the BioSystems® Glycerol phosphate Oxidase / Peroxidase kit.
High-density lipoprotein cholesterol | 7 days
  Change from baseline, using the BioSystems® Direct / Detergent HDL kit
Low-density lipoprotein cholesterol | 7 days
  Change from baseline, using the BioSystems® Cholesterol Oxidase / Peroxidase kit
Creatinine | 7 days
  Change from baseline, using the BioSystems® kit Modified Jaffe's no deproteinization
Blood pressure | 7 days
  Change from baseline, using an OMRON calibrated electronic digital sphygmomanometer model HEM 907 XL. The patient will remain seated in a chair resting his back on the backrest, with a minimum rest of 5 minutes, The average of 3 measurements such as BP will be taken

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Grover-Páez, PhD, Study Director — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No